CLINICAL TRIAL: NCT05279963
Title: Electroacupuncture for Bladder Pain Syndrome: an Randomized Controlled Trial and Study for Central Mechanism
Brief Title: EA for BPS: an RCT and Study for Central Mechanism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yuanyuan Wu, Attending Chinese medicine doctor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-02-13
Record Dates: First submitted 2022-02-16; First posted 2022-03-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Bladder Pain Syndrome
Keywords: electroacupuncture; Randomized Controlled Trial; multi-modal magnetic resonance imaging
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Electroacupuncture; Amitriptyline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the characteristics of acupuncture, acupuncture manipulators cannot be blinded. Nevertheless, to avoid the subjective bias of researchers and subjects, outcome assessment and statistical analysis will be performed by different researchers blinded to the allocation information. Patients are informed that they will receive one of two effective acupuncture interventions after enrollment, and during the treatment, patients in EA or SA groups will be in separate rooms to avoid communication. The participant' s allocated intervention will not be revealed until the statistical analysis reports are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- medication group (Active Comparator): Participants in the medication group will be merely treated with oral administration of amitriptyline capsule. The dosage of amitriptyline is 25mg bid, for 4 weeks. Any changes in the medications of participants will be recorded on diary cards.
  Interventions: Drug: Amitriptyline
- EA group (Experimental): Patients allocated to this group will receive treatment with electroacupuncture. The location of acupoints will be determined based on the National Standard Nomenclature and Location of Acupoints. Patients will receive a total number of 12 EA sessions, with the frequency of 3 sessions per week for 4 weeks.
  Interventions: Procedure: electroacupuncture
- SA group (Sham Comparator): Patients allocated to this group will receive acupuncture in non-meridian and non-acupoints regions. The needles are shallowly inserted to the subcutaneous area, and acupoints are connected to the EA apparatus without electricity. The frequency, intensity and duration of treatment will be the same as the EA group.
  Interventions: Procedure: sham electroacupuncture

INTERVENTIONS:
Procedure: electroacupuncture — The prespecified acupoints applied here will include bilateral Sanyinjiao(SP6), Shenshu(BL23), Ciliao(BL32), Zhongliao(BL33), Zhibian(BL54) .
  Acupuncture treatment is carried out by acupuncturists who have been well trained. Acupuncture will be performed with disposable and sterile needles in the specification of 0.25 ×40 mm(diameter: 0.25mm; Suzhou Medical Products Factory Co., Ltd, China). Electroacupuncture procedures will be performed with electronic instruments (Hans-100A, Nanjing Jisheng Medical TechnologyCo., Ltd, China). Two paired of acupoints (i.e., two Shenshu(BL23) and two Ciliao(BL32), respectively) are connected to the EA apparatus. Alternating-frequency mode is selected and frequency is 2/100 Hz. EA intensity is determined in accordance with patients' endurance. EA will last for 30 min for each treatment. Patients will receive a total number of 12 EA sessions, with the frequency of 3 sessions per week for 4 weeks.
  Arms: EA group
Drug: Amitriptyline — Participants in the medication group will be merely treated with oral administration of amitriptyline capsule. The dosage of amitriptyline is 25mg bid, for 4 weeks. Any changes in the medications of individual participants will be recorded on diary cards.
  Arms: medication group
Procedure: sham electroacupuncture — In the trunk region, the points are 5 cm away from respective acupoints. In the lower limb region, the point is 3 cm away from Sanyinjiao(SP6). All points will only receive shallow insertion.
  Acupuncture will be performed with disposable and sterile needles in the specification of 0.25 ×40 mm(diameter: 0.25mm; Suzhou Medical Products Factory Co., Ltd, China).The needles are shallowly inserted to the subcutaneous area, and acupoints are connected to the EA apparatus without electricity. The frequency, intensity and duration of treatment will be the same as the electric needle group.
  Arms: SA group

SUMMARY:
This is a randomized controlled and assessor-blinded design trial to evaluate the efficacy and safety of acupuncture for bladder pain syndrome(BPS). All eligible participants will be randomly assigned to the medication group(n=21), EA group(n=42) and SA group(n=21) in a 1:2:1 allocation ratio. Participants will receive 4-week treatments phase followed by a 4-week follow-up phase. Outcomes will be assessed at baseline, during the treatment and at the end of the follow-up. Outcome assessors, data managers and statisticians will be blinded to the group allocation, while acupuncturists and participants will not be blinded for obvious reasons. Besides, fMRI will be used to collect spontaneous electrical activity of the brain of patients. In this trial, the investigators assume that electroacupuncture for BPS, compared to amitriptyline, is instrumental in improving symptoms such as pain, frequent micturition and emotional disorder.

DETAILED DESCRIPTION:
Participants will be primarily recruited from gynecology, urology and acupuncture departments during outpatient service. All patients will be randomly assigned to either the medication group, EA group or SA group via random number table. SAS 9.3 software will be adopted to generate random numbers. The independent clinical research assistant will be responsible for generating random numbers and making random allocation cards, each with its group allocation information and sealed into an opaque envelope, which will not be open until the first treatment. According to the order of enrollment, eligible participants will be randomly assigned into the medication, EA or SA group at 1:2:1 ratio under the allocation in the envelope.

Due to the characteristics of acupuncture, acupuncture manipulators cannot be blinded. Nevertheless, to avoid the subjective bias of researchers and subjects, outcome assessment and statistical analysis will be performed by different researchers blinded to the allocation information. Patients are informed that they will receive one of two effective acupuncture interventions after enrollment, and during the treatment, patients in EA or SA groups will be in separate rooms to avoid communication. Outcome assessors and statisticians will be blind to the group allocations. The participant's allocated intervention will not be revealed until the statistical analysis reports are completed.

Participants in the medication group will be merely treated with oral administration of amitriptyline capsule. The dosage of amitriptyline is 25 mg bid, for 4 weeks. Any changes in the medications of individual participants will be recorded on diary cards.

In EA group, acupuncture treatment is carried out by acupuncturists who have been well trained. Acupuncture will be performed with disposable and sterile needles in the specification of 0.25 ×40 mm(diameter: 0.25 mm; Suzhou Medical Products Factory Co., Ltd, China). Patients are asked to lie in a prone position with whole body relaxed. Both the skin around the selected acupoints and the hand of acupuncturists are routinely disinfected, after insertion, manipulations of twirling, lifting and uniform reinforcing reducing manipulation will be performed on all needles to elicit 'deqi'. The compositional sensation of 'deqi' involves with numbness, soreness, distention, aching and heaviness, which are believed to be an essential component for acupuncture efficacy. Electroacupuncture procedures will be performed with electronic instruments (Hans-100A, Nanjing Jisheng Medical TechnologyCo., Ltd, China). Two paired of acupoints (i.e., two Shenshu(BL23) and two Ciliao(BL32), respectively) are connected to the EA apparatus. Alternating-frequency mode is selected and frequency is 2/100 Hz. EA intensity is determined in accordance with patients' endurance. EA will last for 30 min for each treatment. Patients will receive a total number of 12 EA sessions, with the frequency of 3 sessions per week for 4 weeks.

In SA group, Acupuncture will be conducted by well-trained acupuncturists and performed with disposable and sterile needles in the specification of 0.25×40 mm (diameter: 0.25 mm; Suzhou Medical Products Factory Co., Ltd, China). Patients are asked to lie in a prone position with whole body relaxed. Both the skin around the selected acupoint and the hand of acupuncturists are routinely disinfected. The needles are subcutaneously inserted to non-meridian and non-acupoints regions. SA procedures will be performed with electronic instruments (Hans-100A, Nanjing Jisheng Medical Technology Co., Ltd, China). Two paired of points are connected to the electronic instruments. Alternating-frequency mode is selected and the frequency is 2/100 Hz. Different from the EA group, the apparatus will run without electricity in the SA group. The procedure will last for 30 min. Patients will receive a total number of 12 SA sessions, with the frequency of 3 sessions per week for 4 weeks.

Outcomes, such as Visual analog scale, O'Leary-Sant questionnaire, 24-hour voiding diary, Hamilton Anxiety Scale and Hamilton Depression Scale, will be assessed at baseline, during the treatment and at the end of the follow-up. Outcome assessors, data managers and statisticians will be blinded to the group allocation, while acupuncturists and participants will not be blinded for obvious reasons.

Besides, fMRI will be used to collect spontaneous electrical activity of the brain of patients, and the changes of spontaneous electrical activity of specific brain regions, resting brain functional connectivity and information interaction of multifunctional areas will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤70 years, male or female;
* Must fulfill the first and the second diagnostic criteria;
* 30 mm≤ VAS score ≤80mm;
* Participants can fully understand the study protocol and a written informed consent is signed.

Exclusion Criteria:

* Patients with previous bladder stones or other space-occupying lesions;
* Previous positive urine culture or significant abnormal urine routine;
* Significant organic lesions of genitourinary system and pelvic organs;
* Patients suffer from severe primary diseases such as cardiovascular, cerebrovascular, respiratory, liver and kidney, or patients cannot receive EA treatment due to any reasons;
* People with heart stents and other metallic substances in their bodies;
* Women who are pregnant, planning to become pregnant, breast-feeding or allergic to study drugs;
* Patients have participated in other clinical trials within the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
Changes in VAS score for pain intensity from baseline to 2 weeks, 4 weeks and 8 weeks after randomization. | at baseline(week 0)、week 2、week 4 and week 8
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.

SECONDARY OUTCOMES:
Changes in O'Leary-Sant questionnaire from baseline to 4 weeks, 8 weeks after randomization. | at baseline(week 0)、week 4 and week 8
  O'Leary-Sant questionnaire include interstitial cystitis Inflammation Index (ICSI) and interstitial Cystitis Problems Index (ICPI). Both ICSI and ICPI contain 4 questions. ICSI mainly assesses the severity of symptoms and every item estimation score ranges between 0 and 5. The total score ranges from 0 to 20 and higher scores indicate more severe symptoms. ICPI evaluates the degree of distress to the patient and every item estimation score ranges from 0 to 4. The total score ranges from 0 to 16; higher score represent, the more serious the distress.
24-hour voiding diary | every day during the 4-week treatment phase
  The frequency of urination and the special feeling during the urination will be carefully recorded every day.
Changes in Hamilton Anxiety Scale from baseline to 4 weeks, 8 weeks after randomization. | at baseline(week 0)、week 4 and week 8
  Hamilton Anxiety Scale is represented by 14 items. Every item estimation score ranges between 0 and 4. The total score ranges from 0 to 56. Higher the score, severe the situation. In this scale, score 7-14 indicates mild severity, 15-21 represents mild to moderate severity, 22-28 represents moderate severity, and >28 indicates severe condition.
Changes in Hamilton Depression Scale from baseline to 4 weeks, 8 weeks after randomization. | at baseline(week 0)、week 4 and week 8
  Hamilton Depression Scale is is composed of 17 questions. The total score ranges from 0 to 53. The higher the score, the more depressed the patient. In this scale, score 8-16 indicates mild severity, 17-23 represents mild to moderate severity, and 24-53 refers moderates to severe condition.

OTHER OUTCOMES:
fMRI features for BPS before and after 4-week electroacupuncture treatment. | at week 4
  Using BOLD-fMRI at resting-state and diffusion tensor imaging, altered fMRI features in brain for BPS patients will be identified before and after 4-week electroacupuncture treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Aﬃliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanno PM, Erickson D, Moldwin R, Faraday MM; American Urological Association. Diagnosis and treatment of interstitial cystitis/bladder pain syndrome: AUA guideline amendment. J Urol. 2015 May;193(5):1545-53. doi: 10.1016/j.juro.2015.01.086. Epub 2015 Jan 23. PMID 25623737
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Background] Hanno PM. Re-imagining interstitial cystitis. Urol Clin North Am. 2008 Feb;35(1):91-9; vii. doi: 10.1016/j.ucl.2007.09.011. PMID 18061027
- [Background] Konkle KS, Berry SH, Elliott MN, Hilton L, Suttorp MJ, Clauw DJ, Clemens JQ. Comparison of an interstitial cystitis/bladder pain syndrome clinical cohort with symptomatic community women from the RAND Interstitial Cystitis Epidemiology study. J Urol. 2012 Feb;187(2):508-12. doi: 10.1016/j.juro.2011.10.040. Epub 2011 Dec 15. PMID 22177158
- [Background] Nickel JC, Payne CK, Forrest J, Parsons CL, Wan GJ, Xiao X. The relationship among symptoms, sleep disturbances and quality of life in patients with interstitial cystitis. J Urol. 2009 Jun;181(6):2555-61. doi: 10.1016/j.juro.2009.02.030. Epub 2009 Apr 16. PMID 19375108
- [Background] Ouyang H, Chen JD. Review article: therapeutic roles of acupuncture in functional gastrointestinal disorders. Aliment Pharmacol Ther. 2004 Oct 15;20(8):831-41. doi: 10.1111/j.1365-2036.2004.02196.x. PMID 15479354
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Quinlan-Woodward J, Gode A, Dusek JA, Reinstein AS, Johnson JR, Sendelbach S. Assessing the Impact of Acupuncture on Pain, Nausea, Anxiety, and Coping in Women Undergoing a Mastectomy. Oncol Nurs Forum. 2016 Nov 1;43(6):725-732. doi: 10.1188/16.ONF.725-732. PMID 27768139
- [Background] Tsai SL, Fox LM, Murakami M, Tsung JW. Auricular Acupuncture in Emergency Department Treatment of Acute Pain. Ann Emerg Med. 2016 Nov;68(5):583-585. doi: 10.1016/j.annemergmed.2016.05.006. Epub 2016 Jun 8. PMID 27287548
- [Background] Wu YY, Jiang YL, He XF, Zhao XY, Shao XM, Du JY, Fang JQ. Effects of Electroacupuncture with Dominant Frequency at SP 6 and ST 36 Based on Meridian Theory on Pain-Depression Dyad in Rats. Evid Based Complement Alternat Med. 2015;2015:732845. doi: 10.1155/2015/732845. Epub 2015 Mar 4. PMID 25821498
- [Background] Lv TT, Lv JW, Wang SY, Jiang C, Gu YJ, Liu HR. [Efficacy of electroacupuncture nerve stimulation therapy for interstitial cystitis/bladder pain syndrome]. Zhongguo Zhen Jiu. 2019 May 12;39(5):467-72. doi: 10.13703/j.0255-2930.2019.05.003. Chinese. PMID 31099215
- [Background] Min zhi, Hu Xiquan, Chen Xuelian, et al. Clinical Observation of Electroacupuncture Combined with Bladder Irrigation for Bladder Pain Syndrome.Shanghai Journal of Acupuncture and Moxibustion. 2020; 39(02): 192-195.
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Thompson E. Hamilton Rating Scale for Anxiety (HAM-A). Occup Med (Lond). 2015 Oct;65(7):601. doi: 10.1093/occmed/kqv054. No abstract available. PMID 26370845
- [Background] Carneiro AM, Fernandes F, Moreno RA. Hamilton depression rating scale and montgomery-asberg depression rating scale in depressed and bipolar I patients: psychometric properties in a Brazilian sample. Health Qual Life Outcomes. 2015 Apr 2;13:42. doi: 10.1186/s12955-015-0235-3. PMID 25889742
- [Background] Melzer J, Rostock M, Brignoli R, Keck ME, Saller R. Preliminary data of a HAMD-17 validated symptom scale derived from the ICD-10 to diagnose depression in outpatients. Forsch Komplementmed. 2012;19(4):191-6. doi: 10.1159/000342018. Epub 2012 Aug 20. PMID 22964985
- [Background] El-Hefnawy AS, Soliman HMM, Abd-Elbary SOM, Shereif WI. Long-standing nonulcerative bladder pain syndrome: Impact of Thiele massage on bladder and sexual domains. Low Urin Tract Symptoms. 2020 May;12(2):123-127. doi: 10.1111/luts.12291. Epub 2019 Oct 24. PMID 31647172
- [Background] Huang MC, Hsieh CH, Chang WC, Chang ST, Lee MS. Assessment of treatment outcomes of interstitial cystitis with hydrodistention and bladder training by O'Leary-Sant Interstitial Cystitis Symptom and Problem Indices. Taiwan J Obstet Gynecol. 2018 Oct;57(5):718-721. doi: 10.1016/j.tjog.2018.08.019. PMID 30342658
- [Background] Suskind AM, Berry SH, Ewing BA, Elliott MN, Suttorp MJ, Clemens JQ. The prevalence and overlap of interstitial cystitis/bladder pain syndrome and chronic prostatitis/chronic pelvic pain syndrome in men: results of the RAND Interstitial Cystitis Epidemiology male study. J Urol. 2013 Jan;189(1):141-5. doi: 10.1016/j.juro.2012.08.088. Epub 2012 Nov 16. PMID 23164386
- [Background] McLennan MT. Interstitial cystitis: epidemiology, pathophysiology, and clinical presentation. Obstet Gynecol Clin North Am. 2014 Sep;41(3):385-95. doi: 10.1016/j.ogc.2014.05.004. Epub 2014 Jul 9. PMID 25155120
- [Background] Jhang JF, Kuo HC. Pathomechanism of Interstitial Cystitis/Bladder Pain Syndrome and Mapping the Heterogeneity of Disease. Int Neurourol J. 2016 Nov;20(Suppl 2):S95-104. doi: 10.5213/inj.1632712.356. Epub 2016 Nov 22. PMID 27915472
- [Background] Cox A. Management of interstitial cystitis/bladder pain syndrome. Can Urol Assoc J. 2018 Jun;12(6 Suppl 3):S157-S160. doi: 10.5489/cuaj.5324. No abstract available. PMID 29875041
- [Background] Beckett MK, Elliott MN, Clemens JQ, Ewing B, Berry SH. Consequences of interstitial cystitis/bladder pain symptoms on women's work participation and income: results from a national household sample. J Urol. 2014 Jan;191(1):83-8. doi: 10.1016/j.juro.2013.07.018. Epub 2013 Jul 17. PMID 23872030
- [Background] Huffman MM, Slack A, Hoke M. Bladder Pain Syndrome. Prim Care. 2019 Jun;46(2):213-221. doi: 10.1016/j.pop.2019.02.002. Epub 2019 Apr 1. PMID 31030822
- [Background] Marcu I, Campian EC, Tu FF. Interstitial Cystitis/Bladder Pain Syndrome. Semin Reprod Med. 2018 Mar;36(2):123-135. doi: 10.1055/s-0038-1676089. Epub 2018 Dec 19. PMID 30566978
- [Background] Rapkin AJ, Kames LD. The pain management approach to chronic pelvic pain. J Reprod Med. 1987 May;32(5):323-7. PMID 2439689
- [Background] Sun Y, Liu Y, Liu B, Zhou K, Yue Z, Zhang W, Fu W, Yang J, Li N, He L, Zang Z, Su T, Fang J, Ding Y, Qin Z, Song H, Hu H, Zhao H, Mo Q, Zhou J, Wu J, Liu X, Wang W, Pang R, Chen H, Wang X, Liu Z. Efficacy of Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome : A Randomized Trial. Ann Intern Med. 2021 Oct;174(10):1357-1366. doi: 10.7326/M21-1814. Epub 2021 Aug 17. PMID 34399062
- [Derived] Xu Y, Chen Y, Shi Y, Lu J, Wu Z, Liu Z, Chen Y, Ni W, Ding Q, Dai W, Wu X, Fang J, Wu Y. Electro-Acupuncture for Bladder Pain Syndrome: A Protocol of a Randomized Controlled Trial and Study for Central Mechanism. J Pain Res. 2022 Jul 13;15:1959-1970. doi: 10.2147/JPR.S370751. eCollection 2022. PMID 35860417